CLINICAL TRIAL: NCT01539161
Title: Reveal Chagas: Clinical Evidence of the Implantable Cardiac Monitor in Patients With Chagas Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Extremely low enrollment rate
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Reveal Chagas
Record Dates: First submitted 2012-02-09; First posted 2012-02-27 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Chagas Disease; Heart Diseases
Keywords: Chagas Disease; Chagasic; Reveal XT; Implantable Cardiac Monitor; ICM
MeSH Terms: conditions — Chagas Disease; Heart Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reveal XT plus SOC (Experimental): Standard of care treatment plus the Reveal XT Implantable Cardiac Monitor. Treatment will follow the same schedule of the standard of care arm regarding exam, ECG and Holter every 6 months, and an Echo, Chest X-Ray and Stress test every 12 months. The addition will be device interrogation at every 6 month exam. Participation will last 36 months.
  Interventions: Device: Implantable Cardiac Monitor
- Standard of Care (Active Comparator): Standard of care arm as described by exam, ECG and Holter every 6 months, and an Echo, Chest X-Ray and Stress test every 12 months. Participation will last 36 months.
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Device: Implantable Cardiac Monitor — 9529 Reveal XT Implantable Cardiac Monitor as well as the use of 9539 Reveal XT Patient Assistant.
  Other Names: 9529 Reveal XT; 9539 Reveal XT Patient Assistant
  Arms: Reveal XT plus SOC
Procedure: Standard of Care — Standard of care arm including exam, ECG and Holter every 6 months, and an Echo, Chest X-Ray and Stress test every 12 months.
  Other Names: SOC
  Arms: Standard of Care

SUMMARY:
The study "Reveal Chagas: Clinical Evidence of the Implantable Cardiac Monitor in Patients with Chagas Disease" is a prospective, multicenter, randomized study that is being conducted at several centers in Latin America with commercially available products.

The primary study hypothesis is that patients with implantable cardiac monitors will have a shorter time to the decision to treat for electrical or arrhythmic disorders during the follow-up period.

The geography includes Argentina and Colombia.

DETAILED DESCRIPTION:
The purpose is to study the possible benefit of a superior treatment decision rate for cardiac arrhythmias (brady- and or/ tachyarrhythmias) using an implantable cardiac monitor (ICM) in patients with Chagas Disease diagnosed by serology, who are asymptomatic and/or minimally symptomatic. Patients that meet inclusion criteria of the study will be randomized to standard care or standard care plus ICM.

Approximately half of the patients will receive an ICM. All patients will be followed for 36 months. It is expected that the enrollment phase will last 1 year, and that the total study duration will be 4 years. The study is expected to end in 2017. One hundred and two patients are needed for 95% confidence level and 80% statistical power to be randomized into the study, at approximately 5 centers in Latin America. Patients will be considered enrolled once they have signed the Informed Consent. The following additional parameters will also be collected:

* Recorded arrhythmic events stored within the ICM (bradyarrhythmia and tachyarrhythmia)
* Time duration spent in arrhythmia and incidence of symptomatic arrhythmias in patients with an ICM.
* Clinical data on subject outcomes and changes in heart failure as assessed by heart failure hospitalizations, New York Heart Association class and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Have Chagas disease, confirmed by two serological tests.
* Provide evidence through any of the following diagnosis methods: Rest ECG, 24 hour Holter monitoring, electrophysiological study, stress test or loop monitoring, at least one electrical disorder consistent with sinus bradycardia greater than 45 and lower than 60 bpm, sinus arrest not greater than 2.0 seconds, second degree atrial sinus block, intraventricular conduction disorders such as right branch, left branch or a bifascicular blockage type, first degree A-V blockage, or of type I second degree AV Block without associated bradycardia, atrial and/or ventricular arrhythmias that do NOT constitute an indication for pacemaker implant, ICD or mapping and radio frequency ablation.
* Be asymptomatic or having minimal isolated unspecific symptoms not consistent with cardiac arrest, aborted sudden death, syncope, frequent and recurrent palpitations, cardiac failure, and lower extremity edema.
* Have ejection fraction of left ventricle >35%
* Be able to give his/her written informed consent.
* Subject should be > 21 years old.
* Be able to return for follow-up visits as required.

Exclusion Criteria:

* Class I or II (according to AHA/HRS/ESC guidelines) indication for final implantation of pacemaker, ICD, or cardiac resynchronizer.
* Exhibit extrinsic causes of sinus dysfunction or A-V blockage.
* Exhibit infiltrative myocardial diseases such as tumors or associated valvular defects.
* Suffer any concurrent disease that may limit the follow up or evaluation.
* Suffer aftereffects of cerebral embolism.
* Suffer ablation or isolation of pulmonary veins previous to their inclusion in the study.
* Not being able or willing to comply with the follow-up schedule.
* Have previous lesions of the spinal cord or aftereffects of skull trauma.
* Have a record of epilepsy.
* Receive pharmacological treatment for other diseases that may modify the autonomic function.
* Have a record of myocardial infarction.
* History of alcohol abuse or drug addiction.
* History of emotional instability, unstable psychiatric disorders or are under treatment for such disorders.
* Have previously implanted pacemakers, cardiodefibrillators or CRT systems.
* Are included or intend to participate in another study of devices during the course of this study.
* Have a clinical condition that may limit life expectancy to < 36 months.
* Use of Antiarrhythmic drugs, except Beta Blockers

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To compare the time to the physician's decision to treat for electrical disorders (brady/tachyarrhythmias) between the two randomized groups. | 36 months
  The primary endpoint is time to the first decision to implant a device (IPG, CRT-P, ICD or CRT-D) or prescribe anti-arrhythmic drugs.

SECONDARY OUTCOMES:
Summarize the recorded arrhythmic events stored within the ICM (bradyarrhythmia and tachyarrhythmia. | 36 months
  Compute summary statistics for arrhythmic events recorded during follow-up, whether or not related to symptoms, for all patients in the ICM arm, including the total number, distribution (e.g., minimum, maximum, median, quartiles, and standard deviation), number per patient year, number of patients having events and percentage of patients having events. Summary statistics for bradyarrhythmia and tachyarrhythmia events will also be computed separately.
Compute the time duration spent in arrhythmias for ICM patients. | 36 months
  Compute the total duration each ICM patient spends in, 1) atrial arrhythmias and 2) ventricular arrhythmias during the entire follow-up period, and their corresponding distribution (e.g., minimum, maximum, median, quartiles, standard deviation). Compute the average duration each patient spends in an, 1) atrial arrhythmia event, and 2) a ventricular arrhythmia event, and the corresponding distributions.
Compute the incidence of symptomatic arrhythmias in patients with an ICM | 36 months
  Compute the incidence rate of symptomatic arrhythmias in patients with an ICM, overall, and for bradyarrhythmias and tachyarrhythmias separately.
Compare the time to the physician's decision to treat with components of the composite primary endpoint between randomization arms. | 36 months
  Individually compare the time to the physicians' decision to treat with the following between the two randomization arms:
  * A device of any type (IPG, CRT-P, ICD or CRT-D)
  * A pacemaker (IPG)
  * Anti-arrhythmic drug therapy
  * A defibrillator (ICD or CRT-D) or prescribe anti-arrhythmic drug therapy
Compare the mortality rate between randomization arms. | 36 months
  Compare the mortality rate between randomization arms.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Muratore, MD, Study Chair — Medtronic; Diego Venagas, MD, Principal Investigator — Colombia; Jose Carlos Pachon Mateos, MD, Study Chair — Brazil; Luis Medesani, MD, Principal Investigator — Argentina - Hospital Interzonal Gernal de Agudos "General José de San Martin"
Locations (4):
- Argentina (2):
  - Hospital General de Agudos "Juan Fernandez", Buenos Aires, Buenos Aires F.D.
  - Hospital Interzonal General de Agudos "General José de San Martin", La Plata
- Colombia (2):
  - Fundacion Cardioinfantil, Bogotá
  - Hospital Militar Central, Bogotá